CLINICAL TRIAL: NCT00404508
Title: A Phase II Study of Epigenetic Therapy With Hydralazine and Magnesium Valproate to Overcome Chemotherapy Resistance in Refractory Solid Tumors
Brief Title: A Phase II Study of Epigenetic Therapy to Overcome Chemotherapy Resistance in Refractory Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Cancerología (Other Government)
Collaborators: Psicofarma, S.A. De C.V. (Industry); National Council of Science and Technology, Mexico (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 005/32/DII
Record Dates: First submitted 2006-11-25; First posted 2006-11-28 (Estimated); Last update posted 2006-11-28 (Estimated); Status verified 2006-11

CONDITIONS: Refractory Solid Tumors
Keywords: Hydralazine; Magnesium Valproate; Chemotherapy resistance; Epigenetic therapy
MeSH Terms: interventions — Hydralazine; Valproic Acid

INTERVENTIONS:
Drug: Hydralazine and magnesium valproate

SUMMARY:
Chemotherapy resistance, either innate or acquired requires for its development, expression changes on a large number of genes therefore, it has been hypothesized that epigenetic-mediated changes could be the responsible driving force for chemotherapy resistance. Aberrant DNA methylation and histone deacetylation are the main epigenetic alterations hence, their reversal by inhibitors of DNA methylation and histone deacetylases (HDACs) may overcome resistance in refractory solid tumors.

Patients will be treated with hydralazine and magnesium valproate starting from day -7 until chemotherapy ends which consists on the same pre-study protocol regimen on which patients progressed. Response and toxicity were evaluated. Global DNA methylation and HDAC activity were evaluated in the peripheral blood cells, as well as the plasma levels of valproic acid and hydralazine.

DETAILED DESCRIPTION:
Eligible patients after signing informed consent will undergo study evaluation and acetylation status typing before being treated. Patients will begin treatment (day -7) with a daily dose of a slow-release formulation of hydralazine tablets containing either 182 mg for rapid-acetylators or 83 mg for slow-acetylators and slow-release tablets containing 700mg of magnesium valproate at a dose of 40mg/Kb t.i.d. Both hydralazine and magnesium valproate will be administered from day -7 until the last day of the last chemotherapy cycle. Chemotherapy will initiate at day 1 (after seven days of being taken hydralazine and magnesium valproate) with the same pre-study protocol regimen at which patients showed tumor progression. Toxicity will be evaluated after each course of chemotherapy. Response will be evaluated at the third course of chemotherapy. Promoter of selected genes will be evaluated by methylation-specific PCR in serum DNA before and after 7 days of treatment with hydralazine and valproate.

ELIGIBILITY:
Inclusion Criteria:

* Aged18 years and older.
* Histologically proven malignant solid tumors who were receiving their second, third or fourth line of palliative chemotherapy and who showed at the second or third course progressive disease as their maximum response according to the RECIST criteria or to the IGCG CA125 criteria in case of ovarian cancer patients.
* Measurable disease defined by 1 of the following criteria: Any unidimensional measurable lesion ≥ 10 mm by standard MRI or CT scan for solid tumors; or at least 1 non-measurable lesion that is evaluable by nuclear medicine, tumor markers, or other reliable measures.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2; Absolute leukocyte count (≥4000/mm3), platelets ≥100,000/mm3, hemoglobin ≥9.0 g/dL; total bilirubin, aspartate amino transferase (AST) and alanine amino transferase (ALT) <1.5 the upper normal limit (UNL), creatinine ≤1.2 mg/dL or a calculated creatinine clearance of ≥60 mL/min.
* Life expectancy of more than three months,
* Written informed consent.

Exclusion Criteria:

* History of allergy to hydralazine or valproate.
* Past or present condition of rheumatic disease, central nervous system disease, heart failure from aortic stenosis and postural hypotension as diagnosed by a physician.
* Previous use of the experimental drugs (hydralazine and magnesium valproate)
* Pregnancy or breast-feeding.
* Uncontrolled systemic disease or infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2005-09; Study Completion 2006-10

PRIMARY OUTCOMES:
Clinical benefit (complete response, partial response and stable disease)
Safety

SECONDARY OUTCOMES:
Global DNA methylation
HDAC inhibition
Gene promoter demethylation from serum DNA

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Duenas-Gonzalez, MD PhD, Study Director — National Institute of Cancerologia
Locations (1):
- National Institute of Cancerologia, Mexico City, Tlalpan, Mexico

REFERENCES:
- [Derived] Candelaria M, Gallardo-Rincon D, Arce C, Cetina L, Aguilar-Ponce JL, Arrieta O, Gonzalez-Fierro A, Chavez-Blanco A, de la Cruz-Hernandez E, Camargo MF, Trejo-Becerril C, Perez-Cardenas E, Perez-Plasencia C, Taja-Chayeb L, Wegman-Ostrosky T, Revilla-Vazquez A, Duenas-Gonzalez A. A phase II study of epigenetic therapy with hydralazine and magnesium valproate to overcome chemotherapy resistance in refractory solid tumors. Ann Oncol. 2007 Sep;18(9):1529-38. doi: 10.1093/annonc/mdm204. PMID 17761710